CLINICAL TRIAL: NCT07181252
Title: Comparison of Post-operative Pain in Relation to Working Length Assessment by Electronic Apex Locator and Digital Radiography in Permanent Teeth Among Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Rakhi Issrani, Lecturer, Jouf University
Other Study IDs: LCBE 24-03/41
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pediatric; Radiography
Keywords: Digital radiography; Electronic apex locator; Dentistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EAL group: Working length determination using EAL
  Interventions: Diagnostic Test: Working length of root
- DR group: Working length determination using DR
  Interventions: Diagnostic Test: Working length of root

INTERVENTIONS:
Diagnostic Test: Working length of root — EAL Group: Working length was measured using the Root ZX apex locator (J. Morita Corp., Kyoto, Japan), following the manufacturer's instructions. A #15 K-file was connected to the device and advanced until the display indicated "APEX," confirming the location beyond the apical foramen.
  DR Group: Working length was determined using a #15 K-file inserted 1 mm short of the estimated radiographic apex. A digital periapical radiograph was taken, and the working length was adjusted accordingly. Repeated radiographs were obtained until the file tip was 1 mm short of the radiographic apex.

SUMMARY:
This randomized, double-blind clinical trial was conducted at the College of Dentistry, Jouf University, Kingdom of Saudi Arabia, between August 2024 and February 2025. A total of 130 pediatric patients were recruited from the outpatient department.

DETAILED DESCRIPTION:
Sample Size and Participants The sample size was calculated based on a previous study by Guzel et al. [16], which assessed post-operative pain in relation to different working length determination methods. To detect a 10% difference in mean pain scores with 95% confidence and 80% power, a minimum sample of 124 participants was required. Accounting for a 5-10% attrition rate, the final sample size was increased to 130 (65 in each group).

Inclusion Criteria Children aged 10-15 years. Clinical and radiographic diagnosis of irreversible pulpitis. Absence of systemic disease. Permanent first molars with mature apices. No radiographic evidence of root resorption or periodontal bone loss. Written consent from a parent or legal guardian. Exclusion Criteria Medically compromised or psychologically unfit children. Teeth with periapical lesions on radiographs. Teeth with severely curved or calcified canals. Presence of acute or chronic systemic inflammatory conditions. Randomization and Blinding

Participants were randomly allocated into two groups using the coin-flip method:

EAL group: Working length determination using EAL DR group: Working length determination using DR The participants and the investigator of post-operative pain were blinded to the group allocation. All clinical procedures were carried out by a single experienced endodontist who was not involved in pain assessment.

Clinical Procedure All root canal treatments were completed in a single visit under local anesthesia using 2% lignocaine with 1:80,000 epinephrine. Caries excavation and access cavity preparation were performed using sterilized high- and low-speed burs. Patency was confirmed using a #10 K-file.

EAL Group: Working length was measured using the Root ZX apex locator (J. Morita Corp., Kyoto, Japan), following the manufacturer's instructions. A #15 K-file was connected to the device and advanced until the display indicated "APEX," confirming the location beyond the apical foramen.

DR Group: Working length was determined using a #15 K-file inserted 1 mm short of the estimated radiographic apex. A digital periapical radiograph was taken, and the working length was adjusted accordingly. Repeated radiographs were obtained until the file tip was 1 mm short of the radiographic apex.

Canal instrumentation was performed using ProTaper Universal NiTi rotary instruments (Dentsply Maillefer, Switzerland) in a crown-down technique. After initial coronal flaring with an SX file, canals were shaped using S1 and S2 files, followed by F1-F3 files up to 1 mm short of the working length. Irrigation was performed with 2.5% sodium hypochlorite throughout the procedure. Final obturation was completed using the lateral compaction technique with gutta-percha cones and resin-based sealer, followed by restoration with composite resin.

Pain Assessment Pain was evaluated using a 10-point Visual Analog Scale (VAS), where 0 indicated "no pain" and 10 denoted "worst possible pain." Participants were trained to use the scale pre-operatively and were provided with printed forms to record pain at specific post-operative intervals: 6 hours, 12 hours, 24 hours, 48 hours, and 7 days. Pre-operative pain scores were recorded before starting the procedure. This method has been widely used in pediatric endodontic research for subjective pain evaluation [17].

Statistical Analysis Data was analyzed using Statistical Package for Social Sciences version 22.0 (IBM Corp., Armonk, NY, USA). Descriptive statistics were computed for demographic variables. The Chi-square test was used to compare categorical variables such as incidence of post-operative pain between groups. Independent samples t-test was used to compare mean VAS scores between groups, while paired t-test was used to compare pre- and post-operative scores within each group. One-way ANOVA was employed to assess mean VAS scores across different post-operative time intervals. A p-value ≤0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Children aged 10-15 years. Clinical and radiographic diagnosis of irreversible pulpitis. Absence of systemic disease. Permanent first molars with mature apices. No radiographic evidence of root resorption or periodontal bone loss. Written consent from a parent or legal guardian.

Exclusion Criteria:

Medically compromised or psychologically unfit children. Teeth with periapical lesions on radiographs. Teeth with severely curved or calcified canals. Presence of acute or chronic systemic inflammatory conditions.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Pre- and post-operative pain assessment | 1 year
  Pain was evaluated using a 10-point Visual Analog Scale (VAS), where 0 indicated "no pain" and 10 denoted "worst possible pain." Participants were trained to use the scale pre-operatively and were provided with printed forms to record pain at specific post-operative intervals: 6 hours, 12 hours, 24 hours, 48 hours, and 7 days. Pre-operative pain scores were recorded before starting the procedure. This method has been widely used in pediatric endodontic research for subjective pain evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Jouf University, Sakakah, Al Jawf Region, Saudi Arabia